CLINICAL TRIAL: NCT04125745
Title: Phase 2 Open-Label Study of Safety and Efficacy Trial of CXA-10 in Pulmonary Arterial Hypertension
Brief Title: Oral CXA-10 in Pulmonary Arterial Hypertension
Acronym: PAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: negative study outcome from Complexa's multicenter clinical trial; no safety concerns
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Complexa, Inc. (Industry)
Responsible Party: Principal Investigator, Marc A. Simon, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19010004; P01HL103455 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2019-10-14 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — CXA-10

STUDY DESIGN:
Intervention Model Description: One-arm, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CXA-10 (Experimental): Oral CXA-10 300 mg once daily for 12 weeks
  Interventions: Drug: CXA-10

INTERVENTIONS:
Drug: CXA-10 — Each subject will receive oral CXA-10 at the dose of 300 mg once daily for 12 weeks
  Other Names: 10-nitro-9(E)-octadec-9-enoic acid

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of 12-week oral CXA-10 therapy in subjects with pulmonary arterial hypertension, with additional evaluation on the clinical efficacy of oral CXA-10 on changes in hemodynamics, exercise capacity, cardiovascular function and patient reported outcomes.

DETAILED DESCRIPTION:
This is a single-center, one-arm, open-label proof of concept safety study and a phase 2a proof of efficacy pre- and post-assessment study of oral CXA-10 for the treatment of pulmonary arterial hypertension.

The investigators hypothesize that administration of CXA-10 for 12 weeks will improves exercise capacity, cardiovascular function and health related quality of life in pulmonary arterial hypertension patients with limited toxicity.

Subjects who meet the inclusion criteria and none of the exclusion criteria will be scheduled within 4 weeks of screening to receive oral CXA-10 at the dose of 300 mg once daily followed by 12 weeks of open-label CXA-10 treatment and then a 4-week safety follow-up. Additional follow-up assessments by telephone will occur in between each outpatient clinic visit.

ELIGIBILITY:
INCLUSION CRITERIA

The following criteria will be required on ALL subjects:

* Male or female between 18-80 years of age inclusive at Screening
* Weight ≥ 40 kg or 88 lbs
* Have a WHO Classification of Functional Status Class II or III
* Must meet all of the following hemodynamic criteria by means of a right heart catheterization: mPAP of ≥ 25 mmHg, PVR ≥ 3 wood units, PAWP of ≤ 15 mmHg. A clinical RHC done within 2 months is acceptable to determine eligibility
* Meet all of the following pulmonary function test parameters, completed no more than 12 months before Screening or at screening: forced expiratory volume in one second (FEV1) > 60% of predicted normal and forced vital capacity (FVC) ≥ 60%
* A 6 MWD test of ≥ 100 m and ≤ 600 m at Screening
* Participants enrolled in an exercise program for pulmonary rehabilitation must be in a stable program 1 month prior to Screening and must agree to maintain their current level of rehabilitation throughout the study. If subjects are not enrolled in an exercise training program for pulmonary rehabilitation they cannot enroll during the Screening/Baseline Period or throughout the study
* If receiving 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase inhibitors (i.e., statins) subjects must not have changed their dose < 4 weeks prior to Screening
* If receiving simvastatin-containing products: simvastatin (Zocor), Vytorin, or any other combination therapy containing simvastatin, the subject's simvastatin dose should not exceed 20 mg/day Note: Subjects using a simvastatin product at dose > 20 mg/day may be rescreened if their dose has been adjusted to ≤ 20 mg/day, at least 4 weeks prior to Screening with no dose or regimen changes within 4 weeks prior to Baseline
* Subjects must be receiving one or more of the following previously approved PAH therapies: phosphodiesterase type 5 inhibitors (PDE5), endothelin receptor antagonist (ERA), soluble guanylate cyclase (sGC) stimulator, prostanoids, prostacyclin receptor agonists and must be on stable doses ≥ 3 months) with no dose adjustment within 1 month of Screening
* Ability to provide written informed consent

EXCLUSION CRITERIA

Subjects meeting any of the following exclusion criteria at baseline will be excluded from participating in study:

* Portopulmonary hypertension and pulmonary veno-occlusive diseases
* Congenital heart defects (i.e., atrial septal defects, ventricular septal defects, and patent ductus arteriosus) repaired < 1 year prior to Screening (Group 1 classification of Pulmonary Hypertension)
* Systolic blood pressure > 160 or < 90 mmHg or diastolic blood pressure > 110 mmHg at Screening
* An average QTcF on supine triplicate ECGs at Screening (Visit 1) of > 500 msec Acute myocardial infarction or acute coronary syndrome (ST-Elevation Myocardial Infarction (STEMI), Non STEMI (NSTEMI) and/or unstable angina) within the last 90 days prior to Screening
* Recent cerebrovascular accident/transient ischemic attack (CVA/TIA) within the last 90 days prior to Screening
* Recent hospitalization for left heart failure within the last 90 days prior to Screening
* Clinically significant aortic or mitral valve disease defined as greater than moderate regurgitation or moderate stenosis; pericardial constriction; restrictive or constrictive cardiomyopathy; left ventricular dysfunction (LVEF < 50%); left ventricular outflow obstruction; symptomatic coronary artery disease; autonomic hypotension; or fluid depletion in the opinion of the investigator
* Evidence of a life-threatening cardiac arrhythmias on ECG at Screening as determined by the physician investigator
* Personal or family history of congenital prolonged QTc syndrome or sudden unexpected death due to a cardiac reason
* Receiving intravenous inotropes (e.g. dopamine, dobutamine) within 2 weeks prior to Screening
* History of angina pectoris or other condition that was treated with long or short acting nitrates < 12 weeks of Screening
* The subject has a history of herbal or natural medication use (including fish oil) within 2 weeks or 5 half-lives, whichever is longer, prior to Baseline
* Subject has taken prednisone at doses > 15 mg/day; if immunosuppressive medications are used the dose must be stable within 12 weeks prior to Screening and throughout the study
* The subject is currently taking a drug that may affect the assay measurement of serum creatinine (e.g. cimetidine, Bactrim, Pyridium)
* Newly prescribed drug or increased dose of an existing drug that is known to prolong the QTc interval and has been associated with Torsades de Pointes Note: Stable doses of these drugs are permitted (i.e., subject has received the same dose and regimen for at least 30 days prior to Screening with no anticipated changes to the dose or regimen during the course of the study)
* The subject is currently taking dimethyl fumarate (Tecfidera™)
* Females with a positive urine pregnancy test at Screening or prior to dosing or who are pregnant or breastfeeding or who are trying to conceive
* Recent (within 6 months) history of abusing alcohol or illicit drugs
* History of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years or prostate cancer who is not currently or expected, during the study, to undergo radiation therapy, chemotherapy, and/or surgical intervention, or to initiate hormonal treatment
* Cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, central nervous system or psychiatric disease that, in the opinion of the investigator, may adversely affect the safety of the subject and/or efficacy of the investigational product or severely limit the lifespan of the subject other than the condition being studied
* Clinically significant hyperthyroidism or hypothyroidism not adequately treated
* Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)
* The subject has known hypersensitivity to the CXA-10, the metabolites, or formulation excipients
* The subject has had treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to Screening or plans to participate in an investigational drug study at any time during this study

Subjects who fail inclusion/exclusion criteria may be re-screened once.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Simon, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will make individual participant data (IPD) available through a data sharing agreement. After publication, data will be deposited in all available suitable public access databases for archival purposes.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: Through a data sharing agreement

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CXA-10
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CXA-10
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.0 in 12 Weeks
Description: Numbers of treatment-related adverse events is assessed by CTCAE v4.0
Time Frame: Baseline to 12 Weeks
Measure: Number; unit: Events
Arm/Group | CXA-10
Number analyzed (Participants) | 1
Events | 2

2. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance is Measured at Baseline and 12 Weeks by Right Heart Catheterization
Description: Pulmonary vascular resistance (PVR) will be measured by right heart catheterization; results reported as changed from baseline in Woods units. PVR is calculated as (mean pulmonary artery pressure - pulmonary artery wedge pressure)/cardiac output, where pressures are in units of mm Hg and cardiac output is in units of L/min. Pulmonary hypertension is defined as PVR > 3 Woods units. A negative change implies a decrease in PVR which would be considered an improvement.
Time Frame: Baseline and 12 Weeks
Measure: Number; unit: Woods units
Arm/Group | CXA-10
Number analyzed (Participants) | 1
Woods units | -1.2

3. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure is Measured at Baseline and 12 Weeks by Right Heart Catheterization
Description: Pulmonary Artery mean pressure will be measured by right heart catheterization
Time Frame: Baseline and 12 Weeks
Measure: Number; unit: mm Hg
Arm/Group | CXA-10
Number analyzed (Participants) | 1
mm Hg | -5

4. Secondary Outcome: Change From Baseline in RV Function as Measured by Tricuspid Annular Plane Systolic Excursion (TAPSE) as Assessed by Echocardiograms at 12 Weeks
Description: Change from baseline in RV function as measured by tricuspid annular plane systolic excursion (TAPSE) as assessed by echocardiograms at 12 weeks
Time Frame: at baseline and 12 weeks
Population: Drug and funding withdrawn prior to analysis; data were not collected.
Arm/Group | CXA-10
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes From Baseline in Functional Exercise Capacity by Assessing 6 Minute Walk Distance Test
Description: Change from baseline in 6 minute walk distance at 12 weeks
Time Frame: at baseline and 12 weeks
Measure: Number; unit: meters
Arm/Group | CXA-10
Number analyzed (Participants) | 1
meters | 23.5

6. Secondary Outcome: Change From Baseline in Levels of Serum N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) at 12 Weeks
Description: Blood samples will be collected for NT-proBNP analysis
Time Frame: at Baseline and 12 Weeks
Population: Drug and funding withdrawn; data were not collected
Arm/Group | CXA-10
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Functional Status of Patients as Assessed by New York Heart Association Functional Class
Description: The New York Heart Association Classification of Functional Status of Patients with pulmonary hypertension will be used to classify disease severity in PAH. It places patients in one of four categories based on how much they are limited during physical activity.
  Measure Description: Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath). Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry on any physical activity without discomfort. Symptoms of dyspnea at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: at Baseline and 12 Weeks
Population: Drug and funding withdrawn prior to analysis; data were not collected
Arm/Group | CXA-10
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Daily Physical Activity as Measured by a Accelerometer
Description: Continuous physical activity monitoring will be conducted using a noninvasive accelerometer. The device must be worn for a minimum of 7 days at home prior to receiving the first dose of the study drug and prior to the end of the study drug treatment at week 12.
Time Frame: Baseline and 12 Weeks
Population: Drug and funding withdrawn prior to analysis; data were not collected
Arm/Group | CXA-10
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CXA-10
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CXA-10 (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early due to lack of efficacy based on the negative study outcome from the drug company's multicenter clinical trial. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04125745/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04125745/ICF_001.pdf